CLINICAL TRIAL: NCT03699657
Title: Radiofrequency Ablation Using a Separable Clustered Electrode for the Treatment of Hepatocellular Carcinomas: A Randomized Controlled Trial of a Dual-Switching Monopolar Mode Versus a Single-Switching Monopolar Mode
Brief Title: Dual and Single Switching Monopolar RFA Using Separable Clustered Electrode for Treatment of HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNUH-2014-0279
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: RFA
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA with DSM mode (Active Comparator): RFA is performed in dual switching mode using a separable clustered electrode (Octopus®) and a three-channel dual-generator unit.
  Interventions: Device: DSM; Device: Separable clustered electrodes
- RFA with SSM mode (Active Comparator): RFA is performed in single switching mode using a separable clustered electrode (Octopus®) and a three-channel dual-generator unit.
  Interventions: Device: SSM; Device: Separable clustered electrodes

INTERVENTIONS:
Device: DSM — Monopolar RFA using dual switching mode (DSM)
  Arms: RFA with DSM mode
Device: SSM — Monopolar RFA using single switching mode (SSM)
  Arms: RFA with SSM mode
Device: Separable clustered electrodes — A separable clustered electrode is similar to a clustered electrode, although it differs from a conventional clustered electrode in that each individual electrode is separable.
  Other Names: Octopus®

SUMMARY:
This study was conducted to prospectively compare the efficacy, safety and mid-term outcomes of dual-switching monopolar (DSM) radiofrequency ablation (RFA) with those of conventional single-switching monopolar (SSM) RFA in the treatment of hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Recently, dual switching monopolar RFA (DSM-RFA) was developed to enhance further the efficiency of the single switching monopolar RFA (SSM-RFA) in creating ablation zone; Yoon et al. reported that DSM-RFA allowed significantly greater RF energy delivery to target tissue per given time, and then, created significantly larger ablation zone than the SSM-RFA in ex vivo and in vivo animal experiments. A retrospective comparative study by Choi et al. reported that the DSM-RFA created significantly larger ablation volume than, but seemed to show similar LTP rate to the SSM-RFA. Still, whether the physical differences between SSM-RFA and DSM-RFA translate into better clinical outcomes remains an open question. Regarding that the choice of equipment is an essential factor to consider in planning image-guided tumor ablation procedure, we thought that the prospective comparison between DSM-RFA and the SSM-RFA would be helpful for improving results of RFA.

Therefore, the purpose of this study was to prospectively compare the efficacy, safety and mid-term outcomes of DSM-RFA with those of conventional SSM-RFA in the treatment of HCC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HCC (>= 1.5cm and < 5cm in maximal diameter) according to AASLD guideline or LI-RADS on MDCT or liver MRI within 60 days before RFA
* no history of previous locoregional treatment

Exclusion Criteria:

* more than three HCC nodules
* tumors abutting to the central portal vein or hepatic vein with a diameter > 5 mm
* Child-Pugh class C
* tumors with major vascular invasion
* extrahepatic metastasis
* severe coagulopathy (platelet cell count of less than 50,000 cells/mm3 or INR prolongation of more than 50 %)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Minimum diameter of ablative zone | 7 days after RFA
  Minimum diameter of ablative zone on post-RFA CT or MRI in a mm.

SECONDARY OUTCOMES:
Technical success rate | 1 month
  Technical success on 1 month follow-up imaging after RFA (no residual/progressed tumor)
IDR rate | 24 months after RFA
  Cumulative intrahepatic distant recurrence (IDR) rate over two years after RFA
EM rate | 24 months after RFA
  Cumulative extrahepatic metastasis (EM) rate over two years after RFA
1-year local tumor progression (LTP) | 12 months after RFA
  Comparison of rates of LTP in two groups in a year after RFA
2-year LTP | 24 months after RFA
  Comparison of rates of LTP in two groups in two years after RFA

OTHER OUTCOMES:
Complication | 1 month after RFA
  Description and comparison of the type and incidence of major complication after RFA are assessed according to Society of Interventional Radiology (SIR) grading system in two groups.
Volume of ablative zone | 7 days after RFA
  Volume of ablative zone on post-RFA CT or MRI in a mm3.
Ablation time | 1 day
  RFA procedure time in each patient.
Maximal diameter of ablative zone | 7 days after RFA
  Maximal diameter of ablative zone on post-RFA CT or MRI in a mm.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No